CLINICAL TRIAL: NCT06201039
Title: Continuous Local Anesthetic Wound Infusion to Improve Quality of Recovery Following Ablative Surgery and Neck Dissection: a Randomized Controlled Trial.
Brief Title: Continuous Local-anesthetic Wound Infusion for Neck Dissection
Acronym: CLAWED
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: Sixth Affiliated Hospital, Sun Yat-sen University (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: 2022-091
Record Dates: First submitted 2023-04-03; First posted 2024-01-11 (Actual); Last update posted 2024-01-11 (Actual); Status verified 2024-01

CONDITIONS: Head and Neck Cancer
MeSH Terms: conditions — Head and Neck Neoplasms | interventions — Lidocaine; Saline Solution

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Masking Description: Participants, clinicians, data collectors, outcome adjudicators and data analysts will not have access to details of group assignment.
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- CWI Block (Experimental): Prior to the end of neck dissection and any additional procedures, the bilateral catheter will be placed adjacent to the cervical plexus underneath the internal jugular vein, left in place for 24 hours and removed in a similar way to the Redon drainage by the surgeon.
  The Continuous placebo Wound Infusion (CWI) will start immediately at a speed of 4ml/h containing 0.5% lidocaine hydrochloride + 1:400000 adrenaline.
  • Intervention: Drug: 0.5% lidocaine hydrochloride at 4ml/h.
  Interventions: Drug: 0.5% Lidocaine Hydrochloride
- CWI Placebo (Placebo Comparator): Control Intervention: Patients in the control arm will undergo the CWI procedure as well. The infusion will contain 0.9% normal saline + 1:400000 adrenaline at 4ml/h.
  • Intervention: Drug: 0.9% normal saline at 4ml/h.
  Interventions: Drug: 0.9% Normal Saline

INTERVENTIONS:
Drug: 0.5% Lidocaine Hydrochloride — Prior to the end of neck dissection and any additional procedures, the bilateral catheter will be placed adjacent to the cervical plexus underneath the internal jugular vein, left in place for 24 hours and removed in a similar way to the Redon drainage by the surgeon. The CWI block will start immediately at a speed of 4ml/h containing 0.5% lidocaine hydrochloride + 1:400000 adrenaline.
  Other Names: CWI Block
  Arms: CWI Block
Drug: 0.9% Normal Saline — Prior to the end of neck dissection and any additional procedures, the bilateral catheter will be placed adjacent to the cervical plexus underneath the internal jugular vein, left in place for 72 hours and removed in a similar way to the Redon drainage by the surgeon. The CWI placebo will start immediately at a speed of 4ml/h containing 0.9% normal saline + 1:400000 adrenaline.
  Other Names: CWI Placebo
  Arms: CWI Placebo

SUMMARY:
The goal of this study is to assess the efficacy of continuous local anesthetic wound infusion to improve quality of recovery following ablative surgery and neck dissection.

DETAILED DESCRIPTION:
Bilateral cervical plexus catheters are convenient and safe to place under the direct vision of the surgeons during ablative and neck dissection. The investigators hypothesize that continuous local anesthetic wound infusion to block bilateral cervical plexus will improve quality of recovery following ablative surgery and neck dissection. The primary endpoint is the quality of recovery, which will be assessed using the 15-item quality of recovery questionnaire (QoR-15). Secondary endpoints include numeric pain scale, number and proportion of patients on salvage analgesics, Incidence of phrenic nerve block, Incidence of recurrent laryngeal nerve block, length of post-anesthesia care unit (PACU) stay, length of post-operative hospital stay.

ELIGIBILITY:
Inclusion Criteria:

* Over age 18;
* patients with head and neck cancer Undergoing ablative surgery and neck dissection.

Exclusion Criteria:

* Patient refuse;
* Relatively contraindications: severe heart, liver, or kidney dysfunction, coagulation dysfunction, and local anesthetic allergy history;
* Intervention unlikely to be effective: drug abuse history, receiving other types of nerve block treatment;
* Unlikely to complete the follow-up: alcoholism, planned to replace WeChat and phone within three months; the expected life span less than three months;
* Unable to cooperate with the questionnaire and use the patient-controlled analgesia pump.

Ages: 16 Years to 70 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult, Older Adult
Enrollment: 80 (Estimated)
Dates: Start 2024-03-01 (Estimated); Primary Completion 2025-08-31 (Estimated); Study Completion 2025-12-31 (Estimated)

PRIMARY OUTCOMES:
Quality of Recovery | At 24 hours after surgery
  The primary outcome will be the 15-item quality of recovery questionnaire (QoR-15).

SECONDARY OUTCOMES:
Postoperative salvage analgesics | Up to 72 hours after surgery
  Patients will be asked to complete a daily diary for 72 hours that records their daily postoperative salvage analgesics.
Phrenic nerve block | Up to 72 hours after surgery
  Patients will be asked to complete a daily diary for 72 hours that records their daily dyspnea.
Numeric rating scale (NRS) for pain | Up to 72 hours after surgery
  Patients will be asked to complete a daily diary for 72 hours that records the numeric pain rating scale composed of 0 (no pain at all) to 10 (worst imaginable pain).
Recurrent laryngeal nerve block | Up to 72 hours after surgery
  Patients will be asked to complete a daily diary for 72 hours that records their daily hoarseness.
Quality of Recovery | Up to 72 hours after surgery
  The primary outcome will be the 15-item quality of recovery questionnaire (QoR-15).

OTHER OUTCOMES:
Post-anesthesia care unit (PACU) time | Intraoperative (At the end of surgery)
  Length of PACU stay
Post-operative hospital time | Through study completion, an average of 1 year
  Length of hospital stay

CONTACTS AND LOCATIONS:
Overall Officials: Ruan, Study Director — The Sixth Affiliated Hospital, Sun Yat-sen University

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Hinther A, Nakoneshny SC, Chandarana SP, Matthews TW, Hart R, Schrag C, Matthews J, McKenzie CD, Fick GH, Dort JC. Efficacy of Multimodal Analgesia for Postoperative Pain Management in Head and Neck Cancer Patients. Cancers (Basel). 2021 Mar 12;13(6):1266. doi: 10.3390/cancers13061266. PMID 33809273
- [Background] Gostian M, Loeser J, Albert C, Wolber P, Schwarz D, Grosheva M, Veith S, Goerg C, Balk M, Gostian AO. Postoperative Pain Treatment With Continuous Local Anesthetic Wound Infusion in Patients With Head and Neck Cancer: A Nonrandomized Clinical Trial. JAMA Otolaryngol Head Neck Surg. 2021 Jun 1;147(6):553-560. doi: 10.1001/jamaoto.2021.0327. PMID 33830180
- [Background] van den Beuken-van Everdingen MH, de Rijke JM, Kessels AG, Schouten HC, van Kleef M, Patijn J. Prevalence of pain in patients with cancer: a systematic review of the past 40 years. Ann Oncol. 2007 Sep;18(9):1437-49. doi: 10.1093/annonc/mdm056. Epub 2007 Mar 12. PMID 17355955
- [Background] Wick EC, Grant MC, Wu CL. Postoperative Multimodal Analgesia Pain Management With Nonopioid Analgesics and Techniques: A Review. JAMA Surg. 2017 Jul 1;152(7):691-697. doi: 10.1001/jamasurg.2017.0898. PMID 28564673
- [Background] Kehlet H. Multimodal approach to control postoperative pathophysiology and rehabilitation. Br J Anaesth. 1997 May;78(5):606-17. doi: 10.1093/bja/78.5.606. PMID 9175983
- [Background] McLeod RS, Aarts MA, Chung F, Eskicioglu C, Forbes SS, Conn LG, McCluskey S, McKenzie M, Morningstar B, Nadler A, Okrainec A, Pearsall EA, Sawyer J, Siddique N, Wood T. Development of an Enhanced Recovery After Surgery Guideline and Implementation Strategy Based on the Knowledge-to-action Cycle. Ann Surg. 2015 Dec;262(6):1016-25. doi: 10.1097/SLA.0000000000001067. PMID 25692358
- [Background] Tan M, Law LS, Gan TJ. Optimizing pain management to facilitate Enhanced Recovery After Surgery pathways. Can J Anaesth. 2015 Feb;62(2):203-18. doi: 10.1007/s12630-014-0275-x. Epub 2014 Dec 10. PMID 25501696
- [Background] Ladha KS, Patorno E, Huybrechts KF, Liu J, Rathmell JP, Bateman BT. Variations in the Use of Perioperative Multimodal Analgesic Therapy. Anesthesiology. 2016 Apr;124(4):837-45. doi: 10.1097/ALN.0000000000001034. PMID 26835644
- [Background] Schwenk ES, Grant AE, Torjman MC, McNulty SE, Baratta JL, Viscusi ER. The Efficacy of Peripheral Opioid Antagonists in Opioid-Induced Constipation and Postoperative Ileus: A Systematic Review of the Literature. Reg Anesth Pain Med. 2017 Nov/Dec;42(6):767-777. doi: 10.1097/AAP.0000000000000671. PMID 29016552
- [Background] Dort JC, Farwell DG, Findlay M, Huber GF, Kerr P, Shea-Budgell MA, Simon C, Uppington J, Zygun D, Ljungqvist O, Harris J. Optimal Perioperative Care in Major Head and Neck Cancer Surgery With Free Flap Reconstruction: A Consensus Review and Recommendations From the Enhanced Recovery After Surgery Society. JAMA Otolaryngol Head Neck Surg. 2017 Mar 1;143(3):292-303. doi: 10.1001/jamaoto.2016.2981. PMID 27737447
- [Background] Telford RJ, Stoneham MD. Correct nomenclature of superficial cervical plexus blocks. Br J Anaesth. 2004 May;92(5):775; author reply 775-6. doi: 10.1093/bja/aeh550. No abstract available. PMID 15113770
- [Background] Petrucci E, Cofini V, Pizzi B, Coletta R, Blasetti AG, Necozione S, Fusco P, Marinangeli F. Intermediate Cervical Plexus Block in the Management of Persistent Postoperative Pain Post Carotid Endarterectomy: A Prospective, Randomized, Controlled, Clinical Trial. Pain Physician. 2020 Jun;23(3):237-244. PMID 32517389
- [Background] Bhoi D, Bhatia R, Mohan VK, Thakar A, Kalagara R, Sikka K. Efficacy of Ultrasound-Guided Intermediate Cervical Plexus Block by Anterior Route for Perioperative Analgesia in Robotic Thyroidectomy by Retroauricular Approach: A Case Series. A A Pract. 2021 Aug 12;15(8):e01501. doi: 10.1213/XAA.0000000000001501. PMID 34388135
- [Background] Kim JS, Lee J, Soh EY, Ahn H, Oh SE, Lee JD, Joe HB. Analgesic Effects of Ultrasound-Guided Serratus-Intercostal Plane Block and Ultrasound-Guided Intermediate Cervical Plexus Block After Single-Incision Transaxillary Robotic Thyroidectomy: A Prospective, Randomized, Controlled Trial. Reg Anesth Pain Med. 2016 Sep-Oct;41(5):584-8. doi: 10.1097/AAP.0000000000000430. PMID 27380104
- [Background] Bu XS, Zhang J, Zuo YX. Validation of the Chinese Version of the Quality of Recovery-15 Score and Its Comparison with the Post-Operative Quality Recovery Scale. Patient. 2016 Jun;9(3):251-9. doi: 10.1007/s40271-015-0148-6. PMID 26518201